CLINICAL TRIAL: NCT05895994
Title: A Study on the Efficacy, Safety and Cellular Pharmacokinetics of RD13-02 Cell Injection in Patients With Relapsed or Refractory CD7-positive Hematological Malignancies
Brief Title: Research Development13(RD13)-02 Cell Injection in Patients With Relapsed or Refractory Cluster Of Differentiation 7(CD7)-Positive Hematological Malignancies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: MEI HENG (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, MEI HENG, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD13-02-07
Record Dates: First submitted 2023-02-18; First posted 2023-06-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; Hematologic Neoplasms; Neoplasms by Site; Hematologic Diseases
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Neoplasms by Site; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD13-02 cell infusion (Experimental)
  Interventions: Drug: RD13-02 cell infusion

INTERVENTIONS:
Drug: RD13-02 cell infusion — CAR-T cells

SUMMARY:
This is a single-arm, open-label, single-center, phase I study. The primary objective is to evaluate the safety of CD7 Chimeric Antigen Receptor-T(CAR-T) therapy for patients with CD7-positive relapsed or refractory T-Acute Lymphoblastic Leukemia(ALL)/Lymphoblastic Lymphoma(LBL)/Acute Myelogenous Leukemia(AML), and to evaluate the pharmacokinetics of CD7 CAR-T in patients。

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-70
2. Diagnosis of r/r T-ALL/LBL/AML.
3. CD7 positive expression
4. Bone marrow lymphoblasts ≥5% by morphologic evaluation at screening
5. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min, Serum alanine aminotransferase(ALT)/aspartate aminotransferase(AST) < 3×upper limit of normal, Total bilirubin < 1.5×upper limit of normal or ≤1.5mg/dl
6. Left ventricular ejection fraction ≥ 50% .
7. Baseline oxygen saturation ≥ 92% on room air.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
9. The estimated survival time is more than 3 months.
10. Subjects or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Subjects with concomitant genetic syndromes associated with bone marrow failure states.
2. Isolated extramedullary lesions
3. Subjects with some cardiac conditions will be excluded.
4. With uncontrolled active central nervous system leukemia (CNSL), cerebrospinal fluid grade Central Nervous System3(CNS3).
5. History of traumatic brain injury, consciousness disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic disease, which might compromise the ability of the subject to compliance with the obligations under the protocol.
6. History of malignancy other than non-melanoma skin cancer or carcinoma.
7. Primary immune deficiency.
8. Presence of uncontrolled infections.
9. Subjects with some anticancer therapy before CAR-T infusion will be excluded.
10. Active uncontrolled acute infections.
11. Known history of infection with human immunodeficiency virus (HIV); active or latent hepatitis B, hepatitis C and syphilis.
12. Subjects who are receiving systemic steroid therapy prior to screening.

14.Having received live/attenuated vaccine within 4 weeks prior to screening. 15.History of allergy to any component of the cell therapy product. 16.Pregnant or breastfeeding women 17.Any other issue which, in the opinion of the investigator, would make the subjects ineligible for the study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Evaluate at 4 weeks after CAR-T infusion
  The proportion of patients with complete response (CR) /complete response with incomplete blood cell recovery (CRi)
Overall response rate (ORR) | Evaluate at 8 weeks after CAR-T infusion
  The proportion of patients with complete response (CR) /complete response with incomplete blood cell recovery (CRi)
Overall response rate (ORR) | Evaluate at 12 weeks after CAR-T infusion
  The proportion of patients with complete response (CR) /complete response with incomplete blood cell recovery (CRi)

SECONDARY OUTCOMES:
Objective response rate , ORR | Up to 1 years after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and partial response (PR).
Overall response rate with Minimal Residual Disease (MRD)-negative, MRD-ORR | Up to 1 years after CAR-T infusion
  Proportion of patients achieving CR/CRi who is MRD-negative in bone marrow
Duration of remission (DOR) | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Event-free survival (EFS) | Up to 1 years after CAR-T infusion
  The time from first achieving CR/CRi to relapse or death
The proportion of patients who receive hematopoietic stem cell transplantation | Up to 1 years after CAR-T infusion
  The proportion of subjects who achieved remission after infusion who received Hematopoietic Stem Cell Transplantation (HSCT)
Overall survival (OS) | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No